CLINICAL TRIAL: NCT05689138
Title: SCREENING ORAL AND GUT MICROBES AS A MORE ACCURATE NON-INVASIVE TOOL FOR PANCREATIC CANCER EARLY DETECTION: A POPULATION-BASED CASE-CONTROL STUDY IN CHINA
Brief Title: Using Digestive Microbial Information to Enhance the Early Detection of Pancreatic Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Dai Menghua, Professor, Peking Union Medical College Hospital
Other Study IDs: PUMCH-PCAMicrobe-1
Record Dates: First submitted 2023-01-09; First posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PCA: pancreatic cancer patients
  Interventions: Other: Oral and Fecal Sample Collection
- NC: normal control
  Interventions: Other: Oral and Fecal Sample Collection

INTERVENTIONS:
Other: Oral and Fecal Sample Collection — No interventions

SUMMARY:
Pancreatic cancer (PCA) is a leading death-related cancer. There is an urgent need for accurate, noninvasive diagnostic options in the early detection of pancreatic cancer (PCA), since delayed diagnosis increases the risk of metastasis and recurrence. In this study, by analyzing gut and fecal microbial data among the pancreatic versus healthy populations, we aim to establish an early detection tool to improve PCA detection, and to explore potential diagnostic biomarkers.

ELIGIBILITY:
Inclusion Criteria:

PCA Newly diagnosed pancreatic cancer patients; No symptoms of jaundice; Did not yet receive any treatment

NC Individuals who were undergoing routine screenings or physical examination

Exclusion Criteria:

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Present/ past diagnosis of (a) other malignancy, (b) infectious diseases, (c) oral or digestive diseases, (d) mental psychiatric or neurodegenerative diseases, (e) chronic diseases that may affect the organ function; Have received certain medical examinations or interventions within specific periods, including (a) antibiotics, hormonotherapy, or immunosuppressor in the past three months, (b) digestive tract reconstructive operation in the past three months, (c) Frequent use of a cathartic, antidiarrheal, or therapeutic dose of probiotics throughout the past one month, (d) Change of diet throughout the past one month, (e) local antibiotics usage in 1 week(skin, antibacterial mouth wash) (f) oral or digestive examination in 3 days.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
microbial features by 16s rRNA sequencing | within 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Menghua Dai, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- PUMCH, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided